CLINICAL TRIAL: NCT02132715
Title: KAATSU Training to Enhance Physical Function of Older Adults With Osteoarthritis
Acronym: KAATSU-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400300; 1R21AR065039-01A1 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistance exercise (Active Comparator): Traditional isotonic lower-extremity resistance training
  Interventions: Behavioral: Resistance Exercise
- KAATSU exercise (Experimental): Lower-extremity exercise with blood flow mildly restricted
  Interventions: Behavioral: KAATSU exercise

INTERVENTIONS:
Behavioral: Resistance Exercise
  Arms: Resistance exercise
Behavioral: KAATSU exercise
  Arms: KAATSU exercise

SUMMARY:
As the U.S. population ages and the prevalence of osteoarthritis (OA) among older adults rises, the prevention of OA-associated disability is an important public health priority. Accordingly, efficacious interventions are needed to manage pain and maintain physical function among older adults with OA. Because skeletal muscle weakness is a primary contributory factor to the progression of pain and functional decline among persons with OA, optimal interventions are those capable of improving skeletal muscle strength. High-intensity resistance exercise is the best-known method of improving muscle strength; however high-compressive loads typically induce significant joint pain among persons with OA. Accordingly, current recommendations include the performance of low- or moderate-intensity physical exercise - despite the fact that these training paradigms are sub-optimal for enhancing muscle strength. This application proposes conduct a pilot study to investigate the potential of an innovative training paradigm with potential to stimulate improvements in skeletal muscle strength while utilizing low-intensity loads. This paradigm, known as KAATSU training, involves performing low-intensity exercise while externally-applied compression mildly restricts blood flow to the active skeletal muscle. The overarching objective of the present application is to evaluate the efficacy and feasibility of chronic KAATSU training for the improvement of skeletal muscle strength and physical function among persons aged > 60 years with symptomatic knee OA and mild to moderate physical limitations. Up to 72 participants will be recruited to participate in this three month intervention study. Participants will be randomly assigned to one of two intervention conditions: (1) a standard exercise intervention consisting of center-based, moderate-intensity resistance training, or (2) a KAATSU training program matched for overall workload. This study will provide novel information regarding the therapeutic potential of KAATSU training for improving strength and function as well as attenuating pain among these individuals. The study will also provide critical information regarding the long-term, clinical viability of the paradigm by evaluating participant safety, discomfort, and willingness to continually engage in the KAATSU training program.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older
* Radiographic evidence of osteophytes
* Moderate to severe pain score (41-90 mm) recorded on 100-mm visual analog scale after 50-ft walk
* Bilateral standing anterior-posterior radiograph demonstrating Kellgren and Lawrence grade 2 or 3
* OA of the target knee
* Score ≤ 10 on the Short Physical Performance Battery, as an indicator of physical limitation
* Sedentary lifestyle, defined as <150 min/wk of moderate physical activity as assessed by CHAMPS questionnaire
* Willingness to participate in all study procedures

Exclusion Criteria:

* Failure to provide informed consent;
* Regular participation in resistance exercise training within the past 3 months
* Current involvement in supervised rehabilitation program
* Absolute contraindication(s) to exercise training according to American College of Sports Medicine guidelines
* Diagnosed peripheral vascular disease
* Ankle-brachial index < 0.95
* Resting office systolic blood pressure > 160 mm Hg or < 100 mm Hg
* Diastolic blood pressure > 100 mm Hg
* History or family history of thrombosis
* Resistant hypertension, defined by BP > 140/90 despite use of 3 or more antihypertensive medications
* Severe cardiac disease, including New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest or stroke, use of a cardiac defibrillator, or uncontrolled angina
* Deep venous thrombosis
* Known peripheral neuropathy
* History of rheumatoid arthritis
* Lower limb amputation
* Lives in a nursing home; (persons living in assisted or independent housing will not be excluded)
* Significant cognitive impairment, defined as a known diagnosis of dementia or a Mini-Mental State Examination exam score < 24
* Unable to communicate because of severe hearing loss or speech disorder;
* Severe visual impairment, which would preclude completion of the assessments and/or intervention
* Other significant co-morbid disease that would impair ability to participate in the exercise intervention
* Lives outside of the study site or is planning to move out of the area during the study timeframe
* Simultaneous participation in another intervention trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in isokinetic muscle strength | 6 weeks post-randomization, 12 weeks post-randomization

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery score | 12-weeks post-randomization
Change in self-paced walking speed | 6 weeks-post randomization, 12 weeks post-randomization
Change in Late Life Disability Questionnaire score | 12 weeks post-randomization
Change in Western Ontario and McMaster Osteoarthritis Index score | 12 weeks post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buford, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided